CLINICAL TRIAL: NCT04088071
Title: Real-world Experience of Catheter Ablation for the Treatment of Symptomatic ParoxysmaL and Persistent Atrial Fibrillation Using Novel CARTO Technologies: REAL AF Registry
Brief Title: Real-world Experience of Catheter Ablation for the Treatment of Paroxysmal and Persistent Atrial Fibrillation
Acronym: REAL-AF
Status: Recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RAF
Record Dates: First submitted 2019-08-26; First posted 2019-09-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with atrial fibrillation: Subjects with symptomatic PAF or PsAF who, in the opinion of the investigator, are candidates for ablation for AF, age 18 years or older, and are able and willing to comply with all pre-, post-, and follow-up testing and requirements.
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: Catheter ablation — Ablation RF technologies (e.g., THERMOCOOL SMARTTOUCH®, THERMOCOOL SMARTTOUCH® SF).

SUMMARY:
The primary purpose of this registry is to obtain real-world clinical experience of Paroxysmal (PAF) and Persistent (PsAF) Atrial Fibrillation ablation radiofrequency (RF) technologies. Data from the registry will be used to assess clinical outcomes, including procedural efficiency, safety, and long-term, effectiveness of catheter ablation with novel RF technologies in PAF and PsAF patients.

DETAILED DESCRIPTION:
The REAL AF Registry is an observational, prospective, multi-center, non-randomized registry designed to obtain real-world clinical experience of Paroxysmal and Persistent ablation RF technologies (e.g., THERMOCOOL SMARTTOUCH®, THERMOCOOL SMARTTOUCH® SF). Future new contact force technologies may be included as they become available in the market. Patient assessments will occur at the following time points: 1) pre-ablation, 2) procedure, 3) 10-12 weeks, 4) 6 months (monitor only) and 5) 1 year post ablation.

The objective of this registry is to assess clinical outcomes, including procedural efficiency, safety, long-term, effectiveness of RF ablations in the treatment of patients with Paroxysmal or Persistent atrial fibrillation. The outcomes of the registry are: 1) long term effectiveness defined as freedom from atrial arrhythmia recurrence post 90 day blanking period, and 2) acute and late onset complications.

Sites selected for this registry will already have the following pre and post procedure assessments as part of their standard of care:

Patient assessments at the following time points: (1) pre-ablation or baseline, (2) procedure, (3) 10-12 weeks, (4) 6 months (monitor only) and (5) 1 year post ablation.

Pre ablation/baseline assessment should include: TTE (within 6 months of procedure), CHADS2Vasc, sleep apnea, AAD status, OAC, Medical and Arrhythmia History 10-12 Week Follow-Up Office Visit: Physician evaluation, AAD status, OAC usage, repeat TTE, and Arrhythmia Reoccurrence and Treatment Assessment Monitoring: 96-hour continuous heart rhythm monitor scheduled at 6 months and 12 months post ablation, with an event monitor ordered as needed for symptomatic arrhythmias.

12 Month Follow up Office Visit: Physician evaluation, AF Type, AF Monitoring method, Sleep apnea, Post-procedure arrhythmia treatments, AF related symptoms and QOL improvement, AAD and OAC usage, CHA2DS2VASC and Arrhythmia Reoccurrence and Treatment Assessment

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Paroxysmal (AF episode terminate spontaneously within 7 days) or Persistent (AF sustained beyond 7 days) who, in the opinion of the investigator, are candidates for ablation for AF
* 18 years of age or older
* De Novo ablation procedure unless it is a repeat for a patient whose index procedure is also in the registry
* Able and willing to participate in baseline and follow up evaluations for the full length of the registry
* Willing and able to provide informed consent, if applicable

Exclusion Criteria:

* Enrolled in an investigational drug or device clinical trial, or any trial that dictates the treatment plan
* Long-standing persistent AF (AF greater than one year's duration)
* Having a repeat ablation, unless the subject's index ablation procedure is also included in the registry
* In the opinion of the investigator, any known contraindication to an ablation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of adults age 18 years or older with symptomatic Paroxysmal and Persistent Atrial Fibrillation who are candidates for ablation.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness at 90 days | 90 days
  Freedom from atrial arrhythmia recurrence at 90 days post procedure.
Effectiveness at 12 months | 12 months
  Freedom from atrial arrhythmia recurrence at 12 months post procedure.
Long-term Safety | Post-procedure, 3 months, and 12 months
  Adverse events from post-procedure through the 12-month office visit date

SECONDARY OUTCOMES:
AF recurrence | 12 months
  Recurrence seen during monitoring with Dual/ CRT Pacer or ICD; Event Monitor; LinQ; Holter; EKG; TTE
Post-procedure arrhythmia treatments | 12 months
  Treatments for AF post-procedure
AF related symptoms | 12 months
  Presence of: weakness, fluttering, SOB, fatigue, dizziness, decrease in exercise tolerance, chest pain/pressure, heart racing/palpitations, and other (yes/no)
AAD Usage | 12 months
  Antiarrhythmic drug use (and type) post procedure and 12 months
OAC usage | 12 months
  Oral anticoagulant use at 12 months and drug type
CHA2DS2VASC | 12 months
  An estimation of stroke risk for patients with Atrial Fibrillation. Composite score of: Age (<65= 0; 65-74=1; >75=2) + Sex (Female=1; Male=0) + Congestive Heart Failure (Yes =1; No=0) + Hypertension (Yes= 1; No= 0) + Stroke, Transient Ischemic Attack (TIA) or thromboembolism (Yes=2; No=0) + Vascular Disease (Yes=1; No=0) + Diabetes (Yes=1; No=0). Scores range from 0 to 9, with higher scores indicating greater risk for stroke.
Patient reported outcome | 12 months
  How do you feel now compared to pre-ablation?

CONTACTS AND LOCATIONS:
Locations (66):
- United States (64):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Cardiology Associates of Mobile, Mobile, Alabama
  - Valley Heart Rhythm Specialists, Chandler, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Keck School of Medicine, Los Angeles, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Community Memorial Hospital, Ventura, California
  - University HealthCare Alliance, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Colorado Heart and Vascular, Golden, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - Ascension St. Vincent's, Jacksonville, Florida
  - HCA Florida Mercy Hospital, Miami, Florida
  - Naples Community Hospital, Naples, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Baycare Health System, Winter Haven, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northshore University Health System, Evanston, Illinois
  - Prairie Education and Research, Springfield, Illinois
  - Ascension St. Vincent's Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Norton Heart Specialists, Louisville, Kentucky
  - Baptist Health Louisville, Saint Matthews, Kentucky
  - Maine Medical Center, Portland, Maine
  - Capitol CArdiology, Lanham, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - Sparrow Clinical Research, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - CoxHealth, Springfield, Missouri
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Lovelace Health System, Albuquerque, New Mexico
  - Columbia University Medical Center / NewYork-Presbyterian Hospital (CUMC/NYPH), New York, New York
  - Nuvance Health, Poughkeepsie, New York
  - Mission Hospital, Asheville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Mount Carmel Columbus Cardiology Consultants, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Upstate Cardiology, Greenville, South Carolina
  - Carolina Cardiology Associates and OnSite Clinical Solutions, Rock Hill, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Centra Health, Inc. dba Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Bon Secours St. Marys, Midlothian, Virginia
  - CJW Medical Center, Richmond, Virginia
  - Valley Health, Winchester, Virginia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - MercyHealth, Janesville, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Canada (2):
  - Alberta Health, Edmonton, Alberta
  - Southlake Regional Health Centre, Newmarket, Ontario

REFERENCES:
- [Background] Sharma E, Varley A, Osorio J, Thorne C, Varosy P, Metzl M, Rajendra A, Oza S, Morales G, Magnano A, D'Souza B, Sackett M, Sellers M, Silva J, Silverstein J, Ho J, Hoskins M, Kuk R, Romero J, Zei PC. Procedural Trends in Catheter Ablation of Persistent Atrial Fibrillation: Insights From the Real-AF Registry. Circ Arrhythm Electrophysiol. 2023 Jun;16(6):e011828. doi: 10.1161/CIRCEP.123.011828. Epub 2023 May 31. No abstract available. PMID 37254771
- [Background] Kreidieh O, Varley AL, Romero J, Singh D, Silverstein J, Thosani A, Varosy P, Hebsur S, Godfrey BE, Schrappe G, Justice L, Zei PC, Osorio J. Practice Patterns of Operators Participating in the Real-World Experience of Catheter Ablation for Treatment of Symptomatic Paroxysmal and Persistent Atrial Fibrillation (REAL-AF) Registry. J Interv Card Electrophysiol. 2022 Nov;65(2):429-440. doi: 10.1007/s10840-022-01205-0. Epub 2022 Apr 19. PMID 35438393
- [Background] Varley AL, Kreidieh O, Godfrey BE, Whitmire C, Thorington S, D'Souza B, Kang S, Hebsur S, Ravindran BK, Zishiri E, Gidney B, Sellers MB, Singh D, Salam T, Metzl M, Ro A, Nazari J, Fisher WG, Costea A, Magnano A, Oza S, Morales G, Rajendra A, Silverstein J, Zei PC, Osorio J. A prospective multi-site registry of real-world experience of catheter ablation for treatment of symptomatic paroxysmal and persistent atrial fibrillation (Real-AF): design and objectives. J Interv Card Electrophysiol. 2021 Dec;62(3):487-494. doi: 10.1007/s10840-021-01031-w. Epub 2021 Jul 2. PMID 34212280
- [Result] Osorio J, Miranda-Arboleda AF, Velasco A, Varley AL, Rajendra A, Morales GX, Hoyos C, Matos C, Thorne C, D'Souza B, Silverstein JR, Metzl MD, Hebsur S, Costea AI, Kang S, Sellers M, Singh D, Salam T, Nazari J, Ro AS, Mazer S, Moretta A, Oza SR, Magnano AR, Sackett M, Dukes J, Patel P, Goyal SK, Senn T, Newton D, Romero JE, Zei PC; REAL-AF Investigators. Real-world data of radiofrequency catheter ablation in paroxysmal atrial fibrillation: Short- and long-term clinical outcomes from the prospective multicenter REAL-AF Registry. Heart Rhythm. 2024 Nov;21(11):2083-2091. doi: 10.1016/j.hrthm.2024.04.090. Epub 2024 May 19. PMID 38768839
- [Result] Kreidieh O, Hunter TD, Goyal S, Varley AL, Thorne C, Osorio J, Silverstein J, Varosy P, Metzl M, Leyton-Mange J, Singh D, Rajendra A, Moretta A, Zei PC; Investigators of the REAL AF registry. Predictors of first pass isolation of the pulmonary veins in real world ablations: An analysis of 2671 patients from the REAL-AF registry. J Cardiovasc Electrophysiol. 2024 Mar;35(3):440-450. doi: 10.1111/jce.16190. Epub 2024 Jan 28. PMID 38282445
- [Result] Costea A, Diaz JC, Osorio J, Matos CD, Hoyos C, Goyal S, Te C, D'Souza B, Rastogi M, Lopez-Cabanillas N, Ibanez LC, Thorne C, Varley AL, Zei PC, Sauer WH, Romero JE. 50-W vs 40-W During High-Power Short-Duration Ablation for Paroxysmal Atrial Fibrillation: A Multicenter Prospective Study. JACC Clin Electrophysiol. 2023 Dec;9(12):2573-2583. doi: 10.1016/j.jacep.2023.08.005. Epub 2023 Oct 4. PMID 37804258
- [Result] Osorio J, Zei PC, Diaz JC, Varley AL, Morales GX, Silverstein JR, Oza SR, D'Souza B, Singh D, Moretta A, Metzl MD, Hoyos C, Matos CD, Rivera E, Magnano A, Salam T, Nazari J, Thorne C, Costea A, Thosani A, Rajendra A, Romero JE. High-Frequency Low-Tidal Volume Ventilation Improves Long-Term Outcomes in AF Ablation: A Multicenter Prospective Study. JACC Clin Electrophysiol. 2023 Aug;9(8 Pt 2):1543-1554. doi: 10.1016/j.jacep.2023.05.015. Epub 2023 May 18. PMID 37294263
- [Result] Rajendra A, Osorio J, Diaz JC, Hoyos C, Rivera E, Matos CD, Costea A, Varley AL, Thorne C, Hoskins M, Goyal S, Oza S, Magnano A, D'Souza B, Silverstein J, Metzl M, Zei PC, Romero JE. Performance of the REAL-AF Same-Day Discharge Protocol in Patients Undergoing Catheter Ablation of Atrial Fibrillation. JACC Clin Electrophysiol. 2023 Aug;9(8 Pt 2):1515-1526. doi: 10.1016/j.jacep.2023.04.014. Epub 2023 May 18. PMID 37204358
- [Result] Rajendra A, Hunter TD, Morales GX, Zei P, Boo LM, Varley A, Osorio J. Steerable sheath visualizable under 3D electroanatomical mapping facilitates paroxysmal atrial fibrillation ablation with minimal fluoroscopy. J Interv Card Electrophysiol. 2023 Mar;66(2):381-388. doi: 10.1007/s10840-022-01332-8. Epub 2022 Aug 10. PMID 35947317
- [Result] Osorio J, Varley A, Kreidieh O, Godfrey B, Schrappe G, Rajendra A, Silverstein J, Romero J, Rodriguez D, Morales G, Zei P. High-Frequency, Low-Tidal-Volume Mechanical Ventilation Safely Improves Catheter Stability and Procedural Efficiency During Radiofrequency Ablation of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2022 Apr;15(4):e010722. doi: 10.1161/CIRCEP.121.010722. Epub 2022 Mar 25. No abstract available. PMID 35333095